CLINICAL TRIAL: NCT06965829
Title: Single-arm Phase II Clinical Study of Neoadjuvant Chemoimmnotherapy Combined With Node Sparing Radiotherapy for Clinical T3N+ Locally Advanced Esophageal Cancer
Brief Title: The Effect of Neoadjuvant Chemoimmnotherapy Combined With Node Sparing Radiotherapy for cT3N+ EC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Guo Xufeng, associate chief physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025shchest
Record Dates: First submitted 2025-04-25; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Cancer Stage III
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NCIT combined with node sparing radiotherapy for clinical T3N+ locally advanced esophageal cancer (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Carboplatin and Paclitaxel and Radiation Therapy

INTERVENTIONS:
Drug: Tislelizumab — Neoadjuvant immunotherapy (tislelizumab 200 mg d1, q3w × 2 cycles)
Drug: Carboplatin and Paclitaxel and Radiation Therapy — Neoadjuvant chemotherapy (nad-paclitaxel 260 mg/m2 d1 + carboplatin AUC = 5 d1, q3w × 2 cycles) and node sparing radiotherapy (41.4Gy/23 times: 1.8Gy d1-5, qw × 4-5 cycles)

SUMMARY:
Background The promising therapeutic outcomes of neoadjuvant chemoimmnotherapy in the treatment of locally advanced esophageal squamous cell carcinoma (ESCC) have been confirmed by several phase II clinical trials and have been widely demonstrated in clinical work. However, in clinical practice, there have been cases of obvious tumor invasion, such as poor tumor regression after cT3 stage receiving NCIT, which reflects the insufficient effectiveness of NCIT for large T type tumors. It may be necessary to add radiotherapy to further improve the local control effect of tumors, but also means higher toxicity reactions. Node sparing radiotherapy can reduce it and enhance the effect of NCIT, which has been applied to the treatment of locally advanced rectal cancer. The aim of this study was to analyze the safety and efficacy of neoadjuvant chemoimmnotherapy combined with node sparing radiotherapy for clinical T3N+ locally advanced esophageal cancer (CINSREC Study).

Methods Forty eligible patients with pathologically confirmed thoracic ESCC of clinical T3N1-3M0 stage were allocated to receive neoadjuvant immunotherapy (tislelizumab 200 mg d1, q3w × 2 cycles) plus chemotherapy (nad-paclitaxel 260 mg/m2 d1 + carboplatin AUC = 5 d1, q3w × 2 cycles) and node sparing radiotherapy (41.4Gy/23 times: 1.8Gy d1-5, qw × 4-5 cycles) treatment. The primary endpoint of this study is pathological complete remission rate (pCR). The secondary endpoints include major pathological response rate, 2-year DFS in pCR patients, adverse events, and overall survival.

Discussion This protocol was reviewed and approved by the Ethics Committee of Shanghai Chest Hospital. This is the first prospective clinical trial to investigate the safety and efficacy of neoadjuvant chemoimmnotherapy combined with node sparing radiotherapy for clinical T3N+ locally advanced esophageal cancer. We hypothesize that this therapy could be a promising therapeutic strategy that can provide better prognosis and safety

ELIGIBILITY:
Inclusion criteria

* The patient volunteers agreed to participate in the study, signed a consent form, exhibited good compliance, observed the follow-up procedures, and were willing and able to follow the protocol during the study.
* Esophageal squamous cell carcinoma diagnosed by histopathology;
* The patients have not received any systemic or local treatment for esophageal cancer in the past including radiotherapy, chemotherapy, surgery, etc;
* The patients were evaluated as thoracic esophageal cancer through auxiliary examinations and clinical staging as T3N+M0 (according to AJCC 8th edition of esophageal cancer);
* Expected to achieve R0 resection;
* Age range: 18-75 years old, male or female not limited;
* The Eastern Cooperative Oncology Group (ECOG) performance status (PS) score is 0-1；
* The patients planned to undergo surgical treatment after completion of neoadjuvant therapy;
* The patients had no surgical contraindications;
* The main organ functions of patients were normal, including: a) blood routine examination (no blood components, cell growth factors, white blood boosting drugs, platelet boosting drugs, or anemia correcting drugs were allowed to be used within 14 days before the first use of the study drug); Neutrophil count ≥ 1.5 * 10 ^ 9/L, platelet count ≥ 100 * 10 ^ 9/L, hemoglobin ≥ 90g/L; b) Blood biochemistry test: Total bilirubin ≤ 1.5 * ULN, ALT≤2.5*ULN, AST≤2.5*ULN, Serum creatinine ≤ 1.5 * ULN, or creatinine clearance rate ≥ 50mL/min; c) Coagulation function: International normalized ratio (INR) ≤ 1.5 * ULN, activated partial thromboplastin time (APTT) ≤ 1.5 * ULN; d) Blood sugar: in normal range and/or with diabetes, the blood sugar was controlled in a stable state during treatment;
* Female subjects with fertility should undergo serum or urine pregnancy testing within 72 hours before starting the study drug administration, and the result should be negative. Effective contraceptive measures (such as intrauterine devices, birth control pills, or condoms) should be taken during the trial period and at least 3 months after the last administration; For male participants whose partners were women of childbearing age, effective contraceptive measures should be taken during the trial period and within 3 months after the last dose. Exclusion criteria
* Unresectable factors, including tumor reasons that cannot be removed or surgical contraindications that cannot be removed or those who refuse surgery;
* Patients with supraclavicular lymph node metastasis;
* Poor nutritional status, BMI<18.5Kg/m2; If the patient's nutritional support is corrected before enrollment and evaluated by the principal investigator, enrollment can continue to be considered;
* Those who are known to have a history of allergies to the components of this drug regimen;
* Have received or are currently receiving any of the following treatments in the past; a) Any radiotherapy, chemotherapy, or other anti-tumor drugs targeting tumors; b) Within 2 weeks prior to the first use of the investigational drug, immunosuppressive or systemic hormone therapy was being used to achieve immunosuppressive effects (dose>10mg/day prednisone or equivalent dose); In the absence of active autoimmune diseases, inhalation or topical use of steroids and corticosteroids at doses>10mg/day of prednisone or equivalent doses are allowed as substitutes for adrenal cortex hormones; c) Received attenuated live vaccine within 4 weeks prior to the first use of the investigational drug; d) Having undergone major surgery or suffered severe trauma within 4 weeks prior to the first use of the investigational drug;
* History of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation or allogeneic bone marrow transplantation;
* Clinical symptoms or diseases of the heart that have not been well controlled, including but not limited to: (1) NYHA class II or above heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias that have not been clinically intervened or are still poorly controlled after clinical intervention;
* Within 4 weeks prior to the first use of the investigational drug, there has been a severe infection (CTCAE>grade 2), such as severe pneumonia requiring hospitalization, bacteremia, and infection complications; Baseline chest imaging examination suggests the presence of active pulmonary inflammation, symptoms and signs of infection within 14 days prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, except for prophylactic use of antibiotics;
* Have participated in other drug clinical studies within the first 4 weeks of randomization;
* Subjects who currently have interstitial pneumonia or interstitial lung disease, or have a history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or have other pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia that may interfere with immune related pulmonary toxicity assessment and management, or those whose screening CT shows active pneumonia or severe lung function impairment; Active pulmonary tuberculosis;
* Patients with any active autoimmune disease or a history of autoimmune disease with the possibility of recurrence [including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (patients controlled solely through hormone replacement therapy may be included)]; Patients with skin diseases that do not require systemic treatment, such as leukoplakia, psoriasis, alopecia, patients with type I diabetes that can be controlled by insulin treatment, or patients with asthma history, but have completely alleviated in childhood and do not need any intervention can be included in the group; Asthma patients who require intervention with bronchodilators cannot be included in the study;
* There is active hepatitis B (HBV DNA ≥ 2000IU/mL or 10 ^ 4copies/mL) and hepatitis C (hepatitis C antibody is negative, and HCV RNA is higher than the detection limit of the analytical method);
* Diagnosed with other malignant tumors within 5 years prior to the first use of the investigational drug, unless there is a low-risk metastasis or death risk malignant tumor (5-year survival rate>90%), such as adequately treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma in situ, may be considered for inclusion;
* Pregnant or lactating women;
* According to the researchers' assessment, there are other factors that may lead to forced termination of the study, such as having other serious illnesses (including mental illnesses) that require concurrent treatment, alcohol abuse, drug abuse, family or social factors, which may affect the safety or compliance of the subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate (pCR) | 12 weeks

SECONDARY OUTCOMES:
Major Pathological Response Rate (MPR) | 12 weeks
Overall survival (OS) | 2 years
Disease free survival (DFS) | 2 years
Adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou X, Chen C, Zeng Y, Yang Z, Zhuo Y, Wang Y, Zhang L, Cai X, Guo X. Neoadjuvant Chemoimmunotherapy Combined With Node-Sparing Radiotherapy for Clinical T3N+ Locally Advanced Esophageal Squamous Cell Carcinoma: A Prospective Single-Arm, Phase II Study (CINSREC Trial). Thorac Cancer. 2025 Nov;16(22):e70191. doi: 10.1111/1759-7714.70191. PMID 41255050